CLINICAL TRIAL: NCT04891237
Title: A Randomized, Double-Blinded, Placebo-Controlled, Prospective, Multicenter CT to Evaluate Efficacy and Safety of Subcutaneous Immunotherapy in Subjects With Rhinitis With/Without Mild to Moderate Asthma Sensitized to Olive and Grass Pollen
Brief Title: Efficacy and Safety Evaluation for the Treatment of Allergy Against Grass and Olive Pollen
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Inmunotek S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMV03-SIT-027
Record Dates: First submitted 2021-04-30; First posted 2021-05-18 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Rhinitis, Allergic; Rhinoconjunctivitis; Asthma, Allergic
Keywords: Rhinitis/ Rhinoconjunctivitis; Mild to moderate asthma; Allergy; Grasses; Olea
MeSH Terms: conditions — Rhinitis, Allergic; Asthma; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind, placebo-controlled, multicentre, parallel-group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During the trial, both the investigator and the included subjects will be unaware of the treatment each subject is receiving.
  The person in charge of data analysis will also not know the treatment assigned to each subject until the database has been closed.
  So that neither the subject nor the investigator knows what treatment each subject is receiving, all the trial medication is identical in terms of outer packaging and appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 10,000 MG01 + 10,000 T517 (Experimental): 10,000 TU/mL of MG01 + 10,000 TU/mL of T517 of subcutaneous immunotherapy
  Interventions: Biological: 10,000 MG01 + 10,000 T517
- 30,000 MG01 + 10,000 T517 (Experimental): 30,000 TU/mL of MG01 + 10,000 TU/mL of T517 of subcutaneous immunotherapy
  Interventions: Biological: 30,000 MG01 + 10,000 T517
- Placebo subcutaneous (Placebo Comparator): The same solution and presentation as the active treatment, but without active ingredients.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: 10,000 MG01 + 10,000 T517 — Purified and polymerized with glutaraldehyde allergen extract, from a mixture of grasses (Phleum pratense, Holcus lanatus, Poa pratensis, Festuca pratensis, Lolium perenne and Dactylis glomerata) and Olea (Olea europaea), adsorbed on aluminum hydroxide. The other ingredients are: sodium chloride (0.9%), phenol (0.4%) and water for injections
  Other Names: Grasses and olea 10,000
  Arms: 10,000 MG01 + 10,000 T517
Biological: 30,000 MG01 + 10,000 T517 — Purified and polymerized with glutaraldehyde allergen extract, from a mixture of grasses (Phleum pratense, Holcus lanatus, Poa pratensis, Festuca pratensis, Lolium perenne and Dactylis glomerata) and Olea (Olea europaea), adsorbed on aluminum hydroxide. The other ingredients are: sodium chloride (0.9%), phenol (0.4%) and water for injections
  Other Names: Grasses and olea
  Arms: 30,000 MG01 + 10,000 T517
Other: Placebo — The same solution and presentation as the active treatment, but without active ingredients
  Arms: Placebo subcutaneous

SUMMARY:
Prospective, multicenter, randomized, double-blind, placebo-controlled clinical trial of efficacy and safety with subcutaneous immunotherapy in patients with mild to moderate rhinitis / rhinoconjunctivitis with or without mild to moderate asthma sensitized to grasses and olive

DETAILED DESCRIPTION:
Double blind, multicenter, parallel, placebo controlled study. It includes 180 subjects sensitised to olea and grass pollen with mild to moderate rhinitis / rhinoconjunctivitis with or without mild to moderate asthma, from 12 to 65 years of age. Medication treatment during 1 year. The main outcome: CSMS

ELIGIBILITY:
Inclusion Criteria:

1. Subject who has signed the informed consent.
2. Subjects of both sexes aged between 12 and 65 years.
3. Subjects with confirmed clinical history of inhalational allergy (rhinitis and / or moderate-severe intermittent or persistent rhinoconjunctivitis according to the ARIA classification with or without intermittent or persistent controlled mild-moderate asthma according to the GEMA 5.0 classification caused by grass and olive allergy. The diagnosis of asthma will be valid from 12 months prior to signing the informed consent
4. Subjects with a positive prick test (higher papule diameter ≥ 5 mm) to a standardized extract of pollen from grasses (Phleum pratense, Holcus lanatus, Dactylis glomerata, Poa pratensis, Festuca elatior, Lolium perenne), or one of the components of the mixture and an olive extract.
5. Specific IgE (CAP or Immulite) against a mixture of grasses or against one of the components of the mixture of grasses, preferably Phleum pratense and olive or one of the molecular components of allergenic sources with a value > 3,5 KU / L.
6. Women of childbearing age (from menarche) should submit a urine pregnancy test with a negative result at the time of joining the trial.
7. Women of childbearing potential, and men participating in the trial, should commit to using an appropriate method of contraception. Medically acceptable methods of contraception are intrauterine devices placed at least 3 months in advance, surgical sterilization (for example, tubal ligation), barrier methods, or the use of oral contraceptives.
8. Subjects capable of complying with the dosage regimen.
9. Subjects who have a smartphone to record symptoms and medication.
10. Subjects with a negative prick test to coestational pollens. In the case specific IgE is available, the result should be <3,5 kU/L and without relevant symptomatology
11. Subjects with a negative prick test to other aeroallergens (dust mites, epitheliums and fungus). In the case specific IgE is available, the result should be <3,5 kU/L and without relevant symptomatology

Exclusion Criteria:

1. Subjects polysensitized to other aeroallergens with the exception of epithelia with occasional exposure and symptoms
2. Subjects polysensitized to other aeroallergens with the exception non-seasonal pollens with grasses and olive
3. Subjects who have received prior immunotherapy in the preceding 5 years to any aeroallergens.
4. Subjects in which immunotherapy may be subject to an absolute general contraindication according to the criteria of the Immunotherapy Committee of the Spanish Society of Allergy and Clinical Immunology and the European Allergy and Clinical Immunology Immunotherapy Subcommittee.
5. Subjects with severe or uncontrolled persistent asthma, with an FEV1 <70% with respect to the reference value despite adequate pharmacological treatment at the time of inclusion in the trial. Likewise, subjects with intermittent or persistent rhinitis / rhinoconjunctivitis with severe symptoms in which the suspension of oral or systemic antihistamine treatment is contraindicated.
6. Subjects who have previously presented a serious secondary reaction during the performance of diagnostic skin tests using the prick test.
7. Subjects under treatment with ß-blockers.
8. Clinically unstable subjects at the time of enrolment in the trial (acute asthma exacerbation, respiratory infection, feverish process, acute urticaria, etc.).
9. Subjects with active chronic urticaria, severe dermographism, severe atopic dermatitis, sunburns, active psoriasis with lesions in areas where skin tests will be performed, or a history of hereditary angioedema.
10. Subjects who have any pathology in which the administration of adrenaline is contraindicated (hyperthyroidism, HT, heart disease, etc.).
11. Subjects with some other disease not related to moderate rhinoconjunctivitis or asthma, but of potential severity and that may interfere with treatment and follow-up (epilepsy, psychomotor disorder, uncontrolled diabetes, malformations, multiple operations, kidney disease,).
12. Subjects with autoimmune disease (thyroiditis, lupus, etc.), tumor diseases or with a diagnosis of immunodeficiencies.
13. Subject whose condition prevents him / her from offering cooperation and who has severe psychiatric disorders.
14. Subjects with a known allergy to other investigational drug components other than the allergen.
15. Subjects with diseases of the lower respiratory tract other than asthma such as emphysema or bronchiectasis.
16. Subjects who are direct relatives of the researchers.
17. Pregnant or lactating women.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
CSMS: Combined Symptoms and Medication Score | 12 months
  Overall score of symptoms and medication throughout the trial. The minimum score is cero and maximum six, per day

SECONDARY OUTCOMES:
Medication-free days | 12 months
  Number of days that the subjects need no medication
Symptom-free days | 12 months
  Number of days that the subjects have no symptom
Asthmatic exacerbations | 12 months
  Time elapsed until the first appearance of asthmatic exacerbations
Visual Analogue Scale (VAS) | 12 months
  Visual Analogue Scale in which the subject has to indicate in a straight line of 10cm how he/she feels regarding to his allergy symptoms. Being left side very bad and right side very well
Quality of life rhinitis test | 12 months
  Quality of life rhinitis test (ESPRINT-15)
Quality of life asthma test | 12 months
  Control of asthma by Asthma Control Quality questionnaire
Health resources | 12 months
  For each patient, the number of times that due to allergy symptoms has done the following will be counted:
  Have visited the GP, Have made an unscheduled visit to the specialist, Has gone to the emergency room, Has been hospitalized, Have needed to contact the doctor by phone
Immunological parameters | 12 months
  Analyses of total and specific IgE, specific Ig G4
Security parameters | 12 months
  Global rate and severity of AE per administration and per subject
Adverse Reactions | 12 months
  Local and systemic reactions and any medication administered for the treatment of AR

CONTACTS AND LOCATIONS:
Overall Officials: Irán Sánchez, Study Chair — Private Site
Locations (32):
- Spain (32):
  - Cedt de Tarancón, Tarancón, Cuenca
  - Hospital Universitario Principe de Asturias, Alcalá de Henares, Madrid
  - Centro Médico Iza, Tres Cantos, Madrid
  - Hospital Infanta Elena, Valdemoro, Madrid
  - Hospital Clínico Universitario Virgen de Arrixaca, El Palmar, Murcia
  - Private Practice, Albacete
  - Hospital Ntra. Sra. de Sonsoles, Ávila
  - Clinica Dermatologica Y Alergia, Badajoz
  - Hospital Quironsalud Clideba, Badajoz
  - Hospital Universitario Dexeus, Barcelona
  - Clínica privada Barcelona, Barcelona
  - Hospital General Universitario Ciudad Real, Ciudad Real
  - Hospital Quironsalud Córdoba, Córdoba
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Universitario de Jaén, Jaén
  - Hospital Universitari Santa María, Lleida
  - Private practice, Madrid
  - Hospital Universitario Cruz Roja, Madrid
  - Clínica de Asma y Alergia en Madrid | CLÍNICA OJEDA, Madrid
  - Clínica Subiza, Madrid
  - Hospital Carlos Iii, Madrid
  - Hospital Universitario Rey Juan Carlos, Madrid
  - Hospital Quirónsalud Málaga, Málaga
  - Private Practice, Málaga
  - Private Practice, Murcia
  - Private Practice, Palencia
  - Hospital Universitario Infanta Cristina, Parla
  - Clínica privada Sevilla, Seville
  - Hospital Virgen Del Rocío, Seville
  - Hospital Viamed Santa Ángela de La Cruz, Seville
  - Private Practice, Toledo
  - Hospital Recoletas Felipe Ii, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Subiza J, Feliu A, Subiza JL, Uhlig J, Fernandez-Caldas E. Cluster immunotherapy with a glutaraldehyde-modified mixture of grasses results in an improvement in specific nasal provocation tests in less than 2.5 months of treatment. Clin Exp Allergy. 2008 Jun;38(6):987-94. doi: 10.1111/j.1365-2222.2008.02995.x. Epub 2008 Apr 25. PMID 18445082
- [Background] Klimek L, Uhlig J, Mosges R, Rettig K, Pfaar O. A high polymerized grass pollen extract is efficacious and safe in a randomized double-blind, placebo-controlled study using a novel up-dosing cluster-protocol. Allergy. 2014 Dec;69(12):1629-38. doi: 10.1111/all.12513. Epub 2014 Oct 6. PMID 25130503
- [Background] Guzman-Fulgencio M, Caballero R, Lara B, Mena M, Tejera M, Sastre A, Subiza JL, Fernandez-Caldas E, Casanovas M. Safety of immunotherapy with glutaraldehyde modified allergen extracts in children and adults. Allergol Immunopathol (Madr). 2017 Mar-Apr;45(2):198-207. doi: 10.1016/j.aller.2016.08.008. Epub 2016 Dec 7. PMID 27939406